CLINICAL TRIAL: NCT04444869
Title: Phase II Trial of Definitive Chemoradiation With Elective Nodal Irradiation Dose De-escalation for p16 Positive Squamous Cell Carcinoma of the Oropharynx "ENID"
Brief Title: Testing Less Intensive Radiation With Chemotherapy to Treat Low-risk Patients With HPV-positive Oropharyngeal Cancer
Acronym: ENID
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Gregory Biedermann, Assistant Professor of Clinical Radiology / Radiation Oncologist, University of Missouri-Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017520
Record Dates: First submitted 2020-05-28; First posted 2020-06-24 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Cancer of the Head and Neck; Oropharynx Cancer; HPV Positive Oropharyngeal Squamous Cell Carcinoma; Throat Carcinoma
MeSH Terms: conditions — Head and Neck Neoplasms; Oropharyngeal Neoplasms | interventions — Cisplatin

STUDY DESIGN:
Intervention Model Description: All patients are treated with the same approach.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open label single-arm study (Other): All patients will receive concurrent cisplatin and radiation therapy with radiation dose de-escalation to clinically and radiologically uninvolved lymph nodes.
  Interventions: Drug: Cisplatin injection

INTERVENTIONS:
Drug: Cisplatin injection — Standard dose cisplatin given concurrently with radiation therapy

SUMMARY:
This trial will explore giving standard dose chemotherapy and radiation therapy to sites of disease including all lymph nodes involved with HPV-positive oropharyngeal cancer, but administer lower doses of radiation therapy to the lymph nodes that are not known to be involved with cancer. By doing so, it is hypothesized that there will be equally good long term loco-regional and distant disease control but will reduced long term treatment side effects and improved quality of life in persons living well beyond their cancer treatment.

DETAILED DESCRIPTION:
This is a trial of definitive chemotherapy and radiation therapy in human papilloma virus positive oropharyngeal cancers, in a population whose cancer is thought to be highly radio-sensitive. This is a population whose outcomes are already known to be very good with high rates of local and distant control of the disease. With the long term disease control and survival of patients with this disease, long term treatment toxicity and resulting reduction in quality of life poses new problems. This has lead to several studies to examine the role of radiation dose de-escalation through various strategies in attempt to reduce long term toxicity from treatment and yet achieve equivalent long term disease control.

This trial specifically hypothesizes that a lower dose of radiation therapy to the clinically and radiographically uninvolved lymph nodes will no detrimental effect on loco-regional control or overall survival and will improve the long-term side effect profile, particularly with regards to xerostomia and dysphagia. The goal of this study is therefore to determine whether a lower dose to the clinically and radiographically uninvolved lymph nodes can be done safely and with better long-term toxicity profile and better overall quality of life without compromising the expected outcomes of progression free survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients generally must have the psychological ability and general health that permits completion of the study requirements and required follow up.
* Women of childbearing potential and men who are sexually active should be willing and able to use medically acceptable forms of contraception throughout the treatment phase of the trial and until at least 60 days following the last study treatment.
* Pathologically (histologically or cytologically) proven diagnosis of squamous cell carcinoma (including the histological variants papillary squamous cell carcinoma and basaloid squamous cell carcinoma) of the oropharynx (tonsil, base of tongue, soft palate, or oropharyngeal walls); cytologic diagnosis from a cervical lymph node is sufficient in the presence of clinical evidence of a primary tumor in the oropharynx. Clinical evidence should be documented, may consist of palpation, imaging, or endoscopic evaluation, and should be sufficient to estimate the size of the primary (for T stage).
* Patients must have clinically or radiographically evident measurable disease at the primary site or at nodal stations. Tonsillectomy or local excision of the primary without removal of nodal disease is permitted, as is excision removing gross nodal disease but with intact primary site. Limited neck dissections retrieving ≤ 4 nodes are permitted and considered as non-therapeutic nodal excisions.
* Immunohistochemical staining for p16 must be performed on tissue and documented in the pathology report(s) with reported result positive for p16.
* Clinical stage T1-T3, N0-N2c (AJCC, 7th ed.), which is equal to T1-T3, N0-2 (AJCC, 8th ed.) including no distant metastases based on the following diagnostic workup:

  * General history and physical examination within 30 days prior to registration;
  * Fiberoptic exam with laryngopharyngoscopy (mirror and/or fiberoptic and/or direct procedure) within 60 days prior to registration;
  * One of the following combinations of imaging is required within 45 days prior to registration:

    1. A CT scan of the neck (with contrast) and a chest CT scan (with or without contrast);
    2. or an MRI of the neck (with contrast) and a chest CT scan (with or without contrast);
    3. or a CT scan of neck (with contrast) and a PET/CT of neck and chest (with or without contrast);
    4. or an MRI of the neck (with contrast) and a PET/CT of neck and chest (with or without contrast).

Note: A CT scan of neck and/or a PET/CT performed for the purposes of radiation planning may serve as both staging and planning tools.

* Patients will be asked about their personal smoking history prior to enrollment. Only active smokers with greater than 10 pack years will be excluded from the trial. The total number of pack years will be collected at baseline. Current smokers who wish to discontinue will be offered smoking cessation information, and if they are able to discontinue smoking prior to initiation of radiation therapy, they can remain eligible for the trial.

Number of pack-years = [Frequency of smoking (number of cigarettes per day) × duration of cigarette smoking (years)] / 20 Note: Twenty cigarettes is considered equivalent to one pack. The effect of non-cigarette tobacco products on the survival of patients with p16-positive oropharyngeal cancers is undefined.

* Zubrod Performance Status of 0-1 within 30 days prior to registration;
* Adequate hematologic function within 14 days prior to registration, defined as follows:

  * Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3;
  * Platelets ≥ 100,000 cells/mm3;
  * Hemoglobin ≥ 8.0 g/dl; Note: The use of transfusion or other intervention to achieve Hgb ≥ 8.0 g/dl is acceptable.
* Adequate renal function within 14 days prior to registration, defined as follows:

  * Serum creatinine < 1.5 mg/dl or creatinine clearance (CC) ≥ 50 ml/min
* Adequate hepatic function within 14 days prior to registration defined as follows:

  * Bilirubin < 2 mg/dl;
  * AST or ALT < 3 x the upper limit of normal.
* Negative serum pregnancy test within 14 days prior to registration for women of childbearing potential

Exclusion Criteria:

* Cancers considered to be from an oral cavity site (oral tongue, floor mouth, alveolar ridge, buccal or lip), or the nasopharynx, hypopharynx, or larynx, even if p16 positive;
* Carcinoma of the neck of unknown primary site origin (even if p16 positive);
* T1-T2 N0-1 lateralized squamous cell carcinoma of the tonsil.
* Radiographically matted nodes, that span 6 cm or more; N3 disease
* Supraclavicular nodes, defined as nodes visualized on the same axial imaging slice as the clavicle;
* Definitive clinical or radiologic evidence of metastatic disease or adenopathy below the clavicles;
* Gross total excision of both primary and nodal disease; this includes tonsillectomy, local excision of primary site, and nodal excision that removes all clinically and radiographically evident disease.
* Simultaneous primary cancers or separate bilateral primary tumor sites;
* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 5 years (for example, carcinoma in situ of the breast, oral cavity, or cervix are all permissible);
* Prior systemic chemotherapy for the study cancer; note that prior chemotherapy for a different cancer is allowable;
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields;
* Severe, active co-morbidity defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months;
  * Transmural myocardial infarction within the last 6 months;
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration;
  * Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days of registration;
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; note, however, that laboratory tests for liver function and coagulation parameters are not required for entry into this protocol other than those requested in Section 3.2.11 of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2020-09-28 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Rate of PEG tube placement | During the procedure
  To determine rate of PEG tube placement

SECONDARY OUTCOMES:
Progression-free survival | Two years post treatment
  Progression-free survival of 85% or more at measured a 2 years post treatment
Dysphagia index | Baseline, 1 month and 6 months after treatment
  To report the change in dysphagia using the M. D. Anderson Dysphagia Inventory (MDADI) scores. Scores are 0 (lowest functioning) to 100 (highest functioning).
Patient Reported Outcomes | Baseline and 1, 6, and 12 months after end of treatment
  European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire
Survival | At 6 months and at 2 years
  To determine overall survival and progression-free survival
Toxicity profiles | 1 year and 2 years post treatment
  Incidence of Common Terminology Criteria for Adverse Events (CTCAE) grade 2 or higher for mucositis, dysphagia, xerostomia and altered taste
Hypothyroidism incidence | At 1 and 2 years post treatment
  To monitor rate of hypothyroidism

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Biedermann, MD, Principal Investigator — University of Missouri - Ellis Fischel Cancer Center
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No